CLINICAL TRIAL: NCT02940340
Title: Evaluation of Systemic Microvascular Endothelial Dysfunction in Patients Presenting With Infective Endocarditis Using the Imaging Method of Cutaneous Laser Speckle Flowmetry
Brief Title: Evaluation of Systemic Microvascular Endothelial Dysfunction in Patients Presenting With Infective Endocarditis
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: NICBrazil
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Infective Endocarditis
Keywords: infective endocarditis; systemic microcirculation
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Infective endocarditis (IE) is a severe clinical condition with a high in-hospital and 5-year mortality. It has a growing incidence, both related to healthcare and possibly to changes in prophylaxis recommendations regarding oral procedures. Though not a new disease, several aspects in its clinical and laboratory diagnosis remain to be better studied and innovated. The evaluation of systemic microvascular disease has proven crucial in the investigation and comprehension of pathophysiology of cardiovascular diseases, as well as a tool for early diagnosis and prediction of complications. Few studies deal with microcirculation in patients with IE, and so far none utilizing speckle contrast imaging and functional capillary density. The present study will contribute to the investigation of microcirculatory changes in IE and possibly to earlier diagnosis of the condition and/or of its severity and complications. The aim of the study is to evaluate the changes in microvascular bed of patients with both acute and subacute endocarditis by speckle contrast imaging and skin video-capillaroscopy.

DETAILED DESCRIPTION:
This is a cohort study that will include adult patients with active definite infective endocarditis by the modified Duke criteria admitted to our center for treatment. A control group of healthy volunteers, paired by sex and age, will be included. The microcirculatory tests will be performed in an undisturbed quiet room with a defined stable temperature (23 ± 1 °C) after a 20-minute rest in the supine position. Functional capillary density (FCD) defined as the number of spontaneously perfused capillaries per square millimeter of skin area will be assessed by video-microscopy system with an epi-illuminated fiber-optic microscope containing a 100-W mercury vapor lamp light source and an M200 objective with a final magnification of 200×. Images will be acquired and saved for posterior off-line analysis using a semi-automatic integrated system (Micro-vision Instruments, Evry, France). The mean capillary density for each patient will be calculated as the arithmetic mean of visible (i.e., spontaneously perfused) capillaries in three contiguous microscopic fields of 1mm2 each. Capillary recruitment (capillary reserve) will be evaluated using post-occlusive reactive hyperemia (PORH) after arm ischemia for 3 min. Microvascular reactivity will be evaluated using an laser speckle contrast imaging (LSCI) system with a laser wavelength of 785 nm (PeriCam PSI system, Perimed, Sweden) in combination with iontophoresis of acetylcholine (ACh), as an endothelium dependent substance, and nitroprusside (endothelium independent) for noninvasive and continuous measurement of cutaneous microvascular perfusion changes (in arbitrary perfusion units, APU).

ELIGIBILITY:
Inclusion Criteria: Endocarditis Diagnostic Criteria -- Duke Criteria

* Major Diagnostic Criteria
* Positive blood culture for typical Infective Endocarditis organisms (strep viridans or bovis, HACEK, staph aureus without other primary site, enterococcus), from 2 separate blood cultures or 2 positive cultures from samples drawn > 12 hours apart, or 3 or a majority of 4 separate cultures of blood (first and last sample drawn 1 hour apart)
* Echocardiogram with oscillating intracardiac mass on valve or supporting structures, in the path of regurgitant jets, or on implanted material in the absence of an alternative anatomic explanation, or abscess, or new partial dehiscence of prosthetic valve or new valvular regurgitation
* Minor Diagnostic Criteria
* Predisposing heart condition or intravenous drug use
* Temp > 38.0° C (100.4° F)
* Vascular phenomena: arterial emboli, pulmonary infarcts, mycotic aneurysms, intracranial bleed, conjunctival hemorrhages, Janeway lesions
* Immunologic phenomena: glomerulonephritis, Osler nodes, Roth spots, rheumatoid factor
* Microbiological evidence: positive blood culture but does not meet a major criterion as noted above or serological evidence of active infection with organism consistent with endocarditis (excluding coag neg staph, and other common contaminants)
* Echocardiographic findings: consistent with endocarditis but do not meet a major criterion as noted above

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with infective endocarditis according to Duke criteria
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
endothelial-dependent and endothelial-independent microvascular reactivity | two years

SECONDARY OUTCOMES:
systemic capillary density | two years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tibirica, MD, PhD, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barcelos A, Lamas C, Tibirica E. Evaluation of microvascular endothelial function in patients with infective endocarditis using laser speckle contrast imaging and skin video-capillaroscopy: research proposal of a case control prospective study. BMC Res Notes. 2017 Jul 28;10(1):342. doi: 10.1186/s13104-017-2660-3. PMID 28754178